CLINICAL TRIAL: NCT03194893
Title: A Multicenter, International, Rollover Study of Alectinib in Patients With Anaplastic Lymphoma Kinase (ALK)-Positive or Rearranged During Transfection (RET)-Positive Cancer
Brief Title: A Rollover Study of Alectinib in Patients With Anaplastic Lymphoma Kinase (ALK)-Positive or Rearranged During Transfection (RET)-Positive Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BO39694; 2017-000207-24 (EudraCT Number)
Record Dates: First submitted 2017-06-20; First posted 2017-06-21 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Neoplasms
Keywords: Non-small cell lung cancer (NSCLC); Anaplastic lymphoma kinase (ALK); Rearranged during transfection (RET); Alectinib; Crizotinib
MeSH Terms: conditions — Neoplasms; Carcinoma, Non-Small-Cell Lung; Multiple Endocrine Neoplasia Type 2a | interventions — alectinib; Crizotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Alectinib (Experimental): Participants will receive alectinib at the same dose and schedule and according to the same administration guidelines as they received at the time of discontinuation from the parent trial.
  Interventions: Drug: Alectinib
- Crizotinib (Experimental): Participants will receive crizotinib at the same dose and schedule and according to the same administration guidelines as they received at the time of discontinuation from the parent trial.
  Interventions: Drug: Crizotinib

INTERVENTIONS:
Drug: Alectinib — Alectinib capsules 600 mg twice a day (BID) orally until no further clinical benefit is to be expected, unacceptable toxicity, availability of commercial supply, withdrawal of consent, or death, whichever occurs first.
  Arms: Alectinib
Drug: Crizotinib — Crizotinib capsules 250 mg BID orally until no further clinical benefit is to be expected, unacceptable toxicity, availability of commercial supply, withdrawal of consent, or death, whichever occurs first.
  Arms: Crizotinib

SUMMARY:
The purpose of this study is to provide continued treatment with alectinib or crizotinib as applicable to participants with ALK- or RET positive cancer who were previously enrolled in any Roche-sponsored alectinib study and who are deriving continued clinical benefit from alectinib or crizotinib in the parent trial at the time of parent trial closure.

ELIGIBILITY:
Inclusion Criteria:

* Participants enrolled in a Roche-sponsored alectinib trial who are experiencing a clinical benefit from alectinib or crizotinib treatment at the time of discontinuation from the parent trial and for whom a switch to commercial supply is not feasible
* Collected study termination data, including efficacy and safety data, as required by the parent study on the electronic Case Report Form (eCRF)
* For women who are not postmenopausal (≥ 12 months of non-therapy-induced amenorrhea) or surgically sterile (absence of ovaries and/or uterus): agreement to remain abstinent or use single or combined contraceptive methods that result in a failure rate of < 1% per year during the treatment period and for at least 3 months after the last dose of study drug
* For men: agreement to remain abstinent or use a contraceptive method that results in a failure rate of < 1% per year during the treatment period and for at least 3 months after the last dose of study drug.

Exclusion Criteria:

* Evidence of lack of clinical benefit in parent trial during the screening phase of this rollover study
* Permanent discontinuation of alectinib or crizotinib for any reason during the parent study or before first dose of study drug in the rollover study
* Evidence of an adverse event for which the parent protocol stipulates permanent discontinuation
* Pregnant or breastfeeding women
* Ongoing serious adverse event that has not resolved to baseline level or Grade ≤1 prior to first dose of study treatment in the rollover study
* Treatment interruption for more than 21 days due to an adverse event since the last administration of alectinib or crizotinib in the parent trial. Any ongoing adverse events that require temporary treatment interruption must be resolved to baseline grade or assessed as stable and not requiring further treatment interruption by the investigator
* Administration of strong/potent cytochrome P450 (CYP) 3A inhibitors or inducers within 14 days prior to the first dose of treatment on this study and while on treatment with crizotinib
* Any psychological, familial, sociological, or geographical condition potentially hampering compliance with the study protocol requirements and/or follow-up procedures; these conditions should be discussed with the participant before trial entry

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-07-05 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Number of Patients with Serious Adverse Events (SAEs), Non-serious Adverse Events (non-SAEs) and Adverse Events of Special Interest | From first dose of study treatment and until the safety follow-up visit (4 weeks after the last dose of study treatment)
  An AE is considered any unfavorable and unintended sign, symptom, or disease associated with use of study drug, whether or not considered related to study drug. Preexisting conditions that worsened during study and laboratory or clinical tests that resulted in a change in treatment or discontinuation from study drug is reported as adverse events. A SAE is any experience that suggests a significant hazard, contraindication, side effect that: results in death, is life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or is medically significant. Adverse events of special interest are cases of potential drug-induced liver injury that include an elevated alanine transaminase (ALT) or aspartate transaminase (AST) in combination with either an elevated bilirubin or clinical jaundice and suspected transmission of an infectious agent by study drug.
Number of Patients With Clinically Significant Laboratory Values as per Protocol for Selected Safety Laboratory Parameters | From first dose of study treatment and until the safety follow-up visit (4 weeks after the last dose of study treatment)
  Selected safety laboratory parameters include alanine transaminase (ALT), aspartate transaminase (AST), total bilirubin, alkaline phosphatase (ALP), and blood creatine phosphokinase (CPK). Any treatment-emergent abnormal laboratory result accompanied by clinical symptoms or leading to a change in study medication or requiring a change in concomitant therapy is considered clinically significant.

SECONDARY OUTCOMES:
Number and Causes of Death Occurring on Study | From first dose of study treatment and until the safety follow-up visit (4 weeks after the last dose of study treatment)
  Once a patient has permanently discontinued study drug and completed the safety follow-up visit, no further survival data will be collected.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (29):
- United States (2):
  - Chao Family Comprehensive Cancer Center, Orange, California
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
- France (8):
  - Centre Francois Baclesse, Caen
  - Centre Georges François Leclerc, Dijon
  - Centre Oscar Lambret, Lille
  - Centre Leon Berard, Lyon
  - Groupe Hospitalier Sud - Hôpital Haut Lévêque, Pessac
  - Hopital Pontchaillou - CHU de Rennes, Rennes
  - CHU de Toulouse - Hôpital Larrey, Toulouse
  - Hopital Robert Schuman, Vantoux
- Hong Kong (2):
  - Queen Mary Hospital, Hong Kong
  - Queen Elizabeth Hospital Department of Clinical Oncology, Kowloon
- Italy (4):
  - Irccs Centro Di Riferimento Oncologico (CRO), Aviano, Friuli Venezia Giulia
  - Azienda Ospedaliera San Camillo Forlanini - Unità Operativa Complessa di Pneumologia Oncologica 1, Rome, Lazio
  - Azienda Ospedaliero-Universitaria Careggi, Florence, Tuscany
  - Azienda Ospedaliera Di Perugia Ospedale s. Maria Della Misericordia, Perugia, Umbria
- Uniwersyteckie Centrum Kliniczne, Gda?sk, Poland
- Russia (3):
  - FSBSI "Russian Oncological Scientific Center n.a. N.N. Blokhin", Moscow, Moscow Oblast
  - University ?linic of headaches, Moscow, Moscow Oblast
  - City Clinical Oncology Hospital, Moscow, Moscow Oblast
- South Korea (2):
  - Seoul National University Hospital, Seoul
  - Samsung Medical Center, Seoul
- Spain (3):
  - Hospital del Mar, Barcelona
  - Hospital Universitari Dexeus - Grupo Quironsalud, Barcelona
  - Hospital Universitario La Paz, Madrid
- Turkey (Türkiye) (4):
  - Adana Ac?badem Hospital Oncology Department, Adana
  - Istanbul Uni Capa Medical Faculty, Istanbul
  - Ege University Medical Faculty, Izmir
  - Hacettepe Uni Medical Faculty Hospital, S?hhiye, Ankara

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing